CLINICAL TRIAL: NCT02572882
Title: A Multi-center Study to Characterize the Gut Microbiome of Individuals With End-stage Renal Disease Treated With Maintenance Hemodialysis, and to Explore Effects of P-inulin on the Gut Microbiome
Brief Title: Gut Microbiome and p-Inulin in Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Brigham and Women's Hospital (Other); George Washington University (Other); Vanderbilt University (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 823162; U01DK099919 (NIH)
Record Dates: First submitted 2015-08-19; First posted 2015-10-09 (Estimated); Results first posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-09

CONDITIONS: End-Stage Renal Disease; Gut Microbiome Dysbiosis
Keywords: hemodialysis; p-inulin; gut microbiome
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This is a sequential trial that included three sequential phases: 1. Pre-treatment phase: 8 weeks during which no treatment was administered 2. p-Inulin phase: 12 weeks during which p-inulin was administered 8g orally twice daily 3. Post-treatment phase: 8 weeks during which no treatment was administered. Eleven of the 13 participants in the p-inulin phase entered the post-treatment phase. The other two withdrew prior to the post-treatment phase.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Other): This is a sequential study in which participants are observed (no intervention) for 8 weeks (pre-treatment), then participants self-administer p-inulin 8g orally twice daily for 12 weeks (treatment phase), and then observed for a final 8 weeks during which no treatment was administered (post-treatment).
  Interventions: Dietary Supplement: p-inulin

INTERVENTIONS:
Dietary Supplement: p-inulin — 12 week self-administered treatment phase

SUMMARY:
The Microbiome trial is a non-randomized, open-label, sequential, multi-center study of p-inulin for patients with hemodialysis-dependent end-stage renal disease.

DETAILED DESCRIPTION:
This primary objective of this exploratory study is to characterize the safety and tolerability of p-inulin (Prebiotin®, provided by JGI Medical) in altering the composition and function of the human gut microbiome, thereby reducing the generation of gut-derived uremic toxins, improving gut barrier function and attenuating systemic inflammation in patients treated with maintenance hemodialysis. The study also aims to assess the feasibility of conducting a full-scale trial of p-inulin. The primary efficacy parameters of the trial will be intra- and inter-participant variability in gut metabolites and bacterial composition. Secondary parameters of interest include tolerability and safety of p-inulin, willingness of hemodialysis patients to enroll in a study requiring repeated collection of stool samples, and participant adherence to agent treatment and specimen collection schedules.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance hemodialysis therapy for end-stage renal disease
* At least 18 years of age
* At least 90 days since hemodialysis initiation
* Self-reported average stool frequency of at least 1 every other day
* For women of childbearing potential, willingness to use a highly effective method of birth control for up to 4 weeks after the last dose of p-inulin.
* Ability to provide consent

Exclusion Criteria:

* Use of prebiotics or probiotics during the past 8 weeks
* Consumption of probiotic yogurt during the past 2 weeks
* Use of antibiotics within the past 8 weeks
* Presence of HIV infection, chronic wound infection, osteomyelitis, or current hemodialysis
* Inflammatory bowel disease, chronic diarrhea, current C. difficile infection
* Cirrhosis or chronic active hepatitis
* Anticipated kidney transplantation, change to peritoneal dialysis, or transfer to another dialysis unit within 9 months
* Expected survival less than 9 months
* Pregnancy, anticipated pregnancy, or breastfeeding
* Incarceration
* Participation in another intervention study
* Severe anemia defined as hemoglobin <9.0 g/dl within the past 4 weeks as documented in the dialysis unit patient record

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dember, MD, Principal Investigator — University of Pennsylvania; J Richard Landis, PhD, Principal Investigator — Perelman School of Medicine at the University of Pennsylvania
Locations (4):
- United States (4):
  - The George Washington University, Washington D.C., District of Columbia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Kidney Research Institute, University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Raj DS, Sohn MB, Charytan DM, Himmelfarb J, Ikizler TA, Mehrotra R, Ramezani A, Regunathan-Shenk R, Hsu JY, Landis JR, Li H, Kimmel PL, Kliger AS, Dember LM; Hemodialysis Novel Therapies Consortium. The Microbiome and p-Inulin in Hemodialysis: A Feasibility Study. Kidney360. 2021 Jan 15;2(3):445-455. doi: 10.34067/KID.0006132020. eCollection 2021 Mar 25. PMID 35369018

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol allowed for enrollment of up to 20 individuals with the goal or having 10 participants complete the first 20 weeks of the study with satisfactory completeness of biosample collection.
Groups:
- Full Study Cohort: This was a sequential study in which participants moved through 3 phases - 8 weeks during which no treatment was administed, 12 weeks during which p-inulin was self-administered orally, 8g twice daily, and another 8 weeks during which no treatment was administered.
Period: Overall Study
Arm/Group | Full Study Cohort
Started | 13
Completed | 11
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Participant received kidney transplant | 1

BASELINE CHARACTERISTICS:
Population: This trial had a sequential design in which participants moved from pre-treatment phase to the treatment phase and then to the post-treatment phaseThe baseline characteristics for the group of 13 participants is shown under pre-treatment phase.
Groups:
- All Participants: This is a sequential study in which participants are observed (no intervention) for 8 weeks (pre-treatment), then participants self-administer p-inulin 8g orally twice daily for 12 weeks (treatment phase), and then observed for a final 8 weeks during which no treatment was administered (post-treatment).
Arm/Group | All Participants
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Within Participant Variability in Microbiome Composition by Treatment Phase
Description: The weighted UniFrac distance was used to compute the distances for each sample. Weighted UniFrac distance uses species abundance information and weights the branch length with abundance difference. Weighted UniFrac distance is most sensitive to detect change in abundant lineages since it uses absolute abundance difference in its definition.
Time Frame: 28 weeks
Population: Two participants withdrew at the beginning of the second phase of the trial. One participant with antibiotic use was not included in the microbiome composition analysis.
Measure: Median (Inter-Quartile Range); unit: weighted unifrac distrance
Groups:
- Full Study Cohort: This study includes three sequential phases: 1. Pre-treatment phase: 8 weeks during which no treatment was administered 2. p-Inulin phase: 12 weeks during which p-inulin was administered 8g orally twice daily 3. Post-treatment phase: 8 weeks during which no treatment was administered
Arm/Group | Full Study Cohort
Number analyzed (Participants) | 10
weighted unifrac distrance
  pre-treatment | 0.165 [0.111 to 0.208]
  treatment | 0.175 [0.129 to 0.228]
  post-treatment | 0.210 [0.129 to 0.266]

2. Primary Outcome: Within Participant Variability in Stool Metabolome by Treatment Phase
Description: The Euclidean distance was used to compute the distances for each sample. The Euclidean distance is defined as the distance between two points.
  Differences between samples were determined on the basis of distances from the initial measurements to account for participant-level differences in initial abundance of microorganisms.
Time Frame: 28 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Euclidean distance
Arm/Group | Full Study Cohort
Number analyzed (Participants) | 10
Euclidean distance
  pre-treatment | 14.49 [11.93 to 18.15]
  treatment | 15.70 [13.37 to 18.32]
  post-treatment | 16.77 [12.92 to 18.12]

3. Primary Outcome: Within Participant Variability in Plasma Metabolome by Treatment Phase
Description: as for outcome 2
Time Frame: 28 weeks (8 weeks pre-treatment, 12 weeks of treatment, 8 weeks post-treatment)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Euclidean distance
Arm/Group | Full Study Cohort
Number analyzed (Participants) | 10
Euclidean distance
  pre-treatment | 9.48 [8.04 to 10.59]
  treatment | 9.47 [8.77 to 10.60]
  post-treatment | 9.72 [8.76 to 11.09]

4. Secondary Outcome: Change in Score of Gastrointestinal Symptom Rating Scale (GSRS) (Safety Outcome)
Description: Gastrointestinal symptoms as measure by the Gastrointestinal Symptom Rating Scale (GSRS). The GSRS total score is the sum of 15 0-3 items where 0 indicates absence and 3 an extreme degree of the symptom. A higher score indicates worse outcome. The minimum score is 0, the maximum score is 45.
Time Frame: GSRS was assessed at Weeks 0, 4, 8, 12, 16, 20, 24 and 28.
Population: Two participants withdrew at the beginning of the second phase of the trial.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Baseline visit, pre-treatment phase
- Week 4: Week 4 Visit, pre-treatment phase
- Week 8: Week 8 visit, pre-treatment phase
- Week 12: Week 12 visit, treatment phase
- Week 16: Week 16 visit, treatment phase
- Week 20: Week 20 visit, treatment phase
- Week 24: Week 24 visit, post-treatment phase
- Week 28: Week 28 visit, post-treatment phase
Arm/Group | Baseline | Week 4 | Week 8 | Week 12 | Week 16 | Week 20 | Week 24 | Week 28
Number analyzed (Participants) | 13 | 13 | 13 | 11 | 11 | 11 | 11 | 11
score on a scale | 5.69 (3.35) | 6.23 (3.65) | 3.68 (5.36) | 4.36 (3.75) | 6.00 (6.47) | 5.27 (5.37) | 3.45 (2.77) | 3.91 (2.59)

5. Secondary Outcome: Number of Participants Who Discontinued Use of P-inulin (Tolerability Outcome)
Description: -Early discontinuation of p-inulin
Time Frame: 12 weeks
Population: This outcome is only relevant during the p-inulin phase.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-treatment: This phase is the 8-week observation period before the p-inulin treatment phase.
- P-inulin: This phase is the 12 week p-inulin treatment phase (8 grams twice daily, oral).
  p-inulin: 12 week self-administered treatment phase
- Post-treatment: This phase is the 8-week observation period after the p-inulin treatment phase.
Arm/Group | Pre-treatment | P-inulin | Post-treatment
Number analyzed (Participants) | 0 | 11 | 0
Participants | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Who Reduce the Dose of P-inulin (Tolerability Outcome)
Description: -Reduction in p-inulin dose
Time Frame: 12 weeks
Population: Three participants reduced their p-inulin dose. This analysis only applies to the 12 week treatment arm.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-treatment Observation Phase; Post-treatment Observation Phase: 8 weeks during which no treatment was administered
- p-Inulin Phase: 12 weeks during which p-inulin was administered 8g orally twice daily
Arm/Group | Pre-treatment Observation Phase | p-Inulin Phase | Post-treatment Observation Phase
Number analyzed (Participants) | 0 | 11 | 0
Participants | 0 | 3 | 0

7. Secondary Outcome: Number of Participants With Adverse Events (Safety Outcome)
Description: -Adverse events per participant related to treatment as coded using the Medical Dictionary for Regulatory Activities (MedDRA) Coding System
Time Frame: 28 weeks
Measure: Number; unit: participants
Groups:
- Pre-treatment Observation Arm; Post-treatment Observation Arm: 8 weeks during which no treatment was administered
- p-Inulin Arm: 12 weeks during which p-inulin was administered 8g orally twice daily
Arm/Group | Pre-treatment Observation Arm | p-Inulin Arm | Post-treatment Observation Arm
Number analyzed (Participants) | 13 | 11 | 11
participants | 1 | 2 | 0

8. Secondary Outcome: Number of Serious Adverse Events (Safety Outcome)
Description: Serious adverse events categorized by body systems, related to treatment as coded using the Medical Dictionary for Regulatory Activities (MedDRA) Coding System
Time Frame: 28 weeks
Population: This is a sequential trial. The 13 participants from the pre-treatment phase moved to the p-inulin phase. Eleven of the 13 participants entered the post-treatment phase. Two participants withdrew prior to the post-treatment phase.
Measure: Number; unit: Serious Adverse Events
Groups:
- Pre-treatment: This arm is the 8-week observation period before the p-inulin treatment phase.
- P-inulin: This arm is the 12 week p-inulin treatment phase (8 grams twice daily, oral).
  p-inulin: 12 week self-administered treatment phase
- Post-treatment: This arm is the 8-week observation period after the p-inulin treatment phase.
Arm/Group | Pre-treatment | P-inulin | Post-treatment
Number analyzed (Participants) | 13 | 11 | 11
Serious Adverse Events | 3 | 0 | 1

9. Secondary Outcome: Rate of Enrollment Refusal (Feasibility Outcome)
Description: Enrollment refusal rate
Time Frame: 1 year
Population: Data not collected
Arm/Group | Pre-treatment Observation Phase | p-Inulin Phase | Post-treatment Observation Phase
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Stool Specimen Collection Proportion - Protocol Adherence (Feasibility Outcome)
Description: Percent of expected completed protocol-specified stool sample collections
Time Frame: 28 weeks
Population: This is a sequential trial. The 13 participants from the pre-treatment phase moved to the p-inulin phase. Eleven of the 13 participants entered the post-treatment phase. Two participants withdrew prior to the post-treatment arm.
Measure: Number; unit: percentage of expected
Arm/Group | Pre-treatment | P-inulin | Post-treatment
Number analyzed (Participants) | 13 | 11 | 11
percentage of expected | 97 | 100 | 97

11. Secondary Outcome: Blood Specimen Collection Proportion - Protocol Adherence (Feasibility Outcome)
Description: Proportion of completed blood sample collections
Time Frame: 28 weeks
Population: as for outcome 8
Measure: Number; unit: percentage of expected
Groups:
- P-inulin: This phase is the 12 week p-inulin treatment phase (8 grams twice daily, oral).
Arm/Group | Pre-treatment | P-inulin | Post-treatment
Number analyzed (Participants) | 13 | 11 | 11
percentage of expected | 99 | 100 | 94

12. Secondary Outcome: Adherence Rate of P-inulin Use (Feasibility Outcome)
Description: Proportion of p-inulin packets used
Time Frame: 12 weeks
Population: as for outcome 8
Measure: Number; unit: percent
Arm/Group | Pre-treatment | P-inulin | Post-treatment
Number analyzed (Participants) | 13 | 11 | 11
percent | 0 | 89.5 | 0

13. Secondary Outcome: Rate of Study Withdrawal (Feasibility Outcome)
Description: Number of withdrawals during each phase of the study
Time Frame: 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-treatment | P-inulin | Post-treatment
Number analyzed (Participants) | 13 | 11 | 11
Participants | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: 28 weeks from Baseline to End of Study
Description: This is a sequential trial. The 13 participants from the pre-treatment phase moved to the p-inulin phase. Eleven of the 13 participants entered the post-treatment phase. Two participants withdrew prior to the post-treatment phase.
Arm/Group | Pre-treatment | P-inulin | Post-treatment
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/13 | 0/11 | 1/11
Other Adverse Events (participants affected / at risk) | 1/13 | 2/11 | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-treatment (N=13) | P-inulin (N=11) | Post-treatment (N=11)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Graft dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-treatment (N=13) | P-inulin (N=11) | Post-treatment (N=11)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT02572882/Prot_SAP_000.pdf
  • Informed Consent Form (2015-09-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT02572882/ICF_001.pdf